CLINICAL TRIAL: NCT04886869
Title: Impact of Caffeine Consumption on Markers of the Autonomic Nervous System
Brief Title: Caffeine and the Autonomic Nervous System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, PD Dr. Stefan Brunner, Prof., LMU Klinikum
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CaffeineLMU
Record Dates: First submitted 2021-04-30; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Autonomic Nervous System Imbalance
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coffee (Experimental): Oral consumption of 3 cups of coffee containing 240 mg caffeine
  Interventions: Dietary Supplement: caffeine
- Energy drink (Experimental): Oral consumption of 750 mL of a commercial energy drink containing 240 mg caffeine
  Interventions: Dietary Supplement: caffeine
- Placebo (Placebo Comparator): Oral consumption of 750 mL water
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — oral consumption

SUMMARY:
Caffeine consumption has been linked to dysfunction of the autonomic nervous system. In this study the investigators analyze the effects of caffeine containing drinks (including energy drinks and coffee) on ECG based parameters of the autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* > 18 years

Exclusion Criteria:

* known cardiovascular disease
* other diseases which may influence the autonomic nervous system
* medication which may influence the autonomic nervous system
* prior caffeine consumption (<24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate (HR) | 2 hours
  ECG-based analysis of heart rate (beats per minute)

SECONDARY OUTCOMES:
Periodic repolarization dynamics (PRD) | 2 hours
  ECG-based analysis of repolarization instability (deg²)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Munich (LMU Klinikum), Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuttler D, Rudi WS, Bauer A, Hamm W, Brunner S. Impact of energy drink versus coffee consumption on periodic repolarization dynamics: an interventional study. Eur J Nutr. 2022 Aug;61(5):2847-2851. doi: 10.1007/s00394-022-02853-8. Epub 2022 Mar 10. PMID 35266046